CLINICAL TRIAL: NCT01710995
Title: A Randomised, Three-Period, Single Dose, Open-Label, Crossover Study to Investigate the Relative Bioavailability and Pharmacodynamic Profiles of a Zegerid 20mg Capsule, Zegerid 20mg Powder for Oral Suspension and Losec 20mg Capsule in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: A Three-Period Study to Investigate the Relative Bioavailability and Pharmacodynamic Profiles of a Zegerid 20mg Capsule, Zegerid 20mg Powder for Oral Suspension and Losec 20mg Capsule in Healthy Adult Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZEG-02/2010 (BE)
Record Dates: First submitted 2012-08-03; First posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Acid Reflux; Gastro Oesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — omeprazole, sodium bicarbonate drug combination; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Zegerid 20mg capsule (Active Comparator): Zegerid 20mg capsule (20mg omeprazole and 1100mg sodium carbonate
  Interventions: Drug: Zegerid
- Zegerid 20mg powder for oral suspension (Active Comparator): Zegerid 20mg powder for oral suspension (20mg omeprazole and 1680mg sodium bicarbonate)
  Interventions: Drug: Zegerid
- Losec 20mg capsule (Active Comparator): Losec 20mg capsule (20mg omeprazole)
  Interventions: Drug: Losec

INTERVENTIONS:
Drug: Zegerid
  Arms: Zegerid 20mg capsule; Zegerid 20mg powder for oral suspension
Drug: Losec
  Arms: Losec 20mg capsule

SUMMARY:
The purpose of this study is to assess the effectiveness of Zegerid 20mg capsules and powder and Losec 20mg capsules in healthy volunteers under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteers aged 18 - 45 years.
* Non-smokers from three months before receiving the first dose and for the duration of the study, confirmed by negative urinary cotinine test at screening and check-in.
* Body mass index (BMI) ≥ 18.0 and ≤ 27.9 kg/m2.
* Able to voluntarily provide written informed consent to participate in the study.
* Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol.
* Able and willing to have a nasogastric tube/probe inserted.
* Females must be post-menopausal (for at least one year and confirmed by serum FSH at screening), surgically sterile, practicing true sexual abstinence or using an acceptable form of effective contraception throughout the study from the following list: contraceptive implants, injectables, oral contraceptives, intrauterine system (IUS), some intrauterine devices (IUDs), vasectomised partner or barrier method (condom or occlusive cap) with spermicidal foam/gel/film/cream/suppository.
* Hormonal and IUD methods of contraception must be established for a period of three months prior to dosing and cannot be changed or altered during the study.
* Females of childbearing potential must have a negative pregnancy test at screening and check-in.
* Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).
* The volunteer's primary care physician must confirm that there is nothing in their medical history that would preclude their enrolment into this clinical study.

Exclusion Criteria:

* Positive for HIV, hepatitis B or hepatitis C.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease as determined by the Investigator.
* History of gastric or duodenal ulcer.
* History of hiatus hernia.
* Significant history of reflux symptoms on clinical judgement.
* Diagnosis of conditions likely to result in a hypersecretory gastric acid state e.g. Zollinger-Ellison Syndrome.
* Positive serology test result for H. pylori at screening.
* Clinically significant deviated nasal septum or other nasopharyngeal obstruction, or inability to tolerate or site a nasogastric tube at screening.
* Hypersensitivity or any other contraindication to Zegerid® or Losec®.
* History or presence of any clinically significant drug allergy.
* Female subjects who are pregnant or lactating.
* Laboratory values at screening which are deemed to be clinically significant as determined by the Investigator.
* Any clinically relevant history of drug or alcohol abuse.
* Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study.
* Participation in a clinical drug study during the 90 days preceding the initial dose of study medication.
* Any significant illness during the screening period preceding the initial dose of study medication.
* Donation of blood or blood products within 90 days prior to study drug administration, or at any time during the study, except as required by this protocol.
* Consumption of alcoholic beverages or xanthine-containing products within 24 hours before confinement or during study confinement.
* Consumption of cruciferous vegetables or chargrilled foods within 48 hours before confinement or during study confinement.
* Consumption of grapefruit or grapefruit juice from seven days before confinement and until the end of the study.
* Use of any prescription or over-the-counter medication (including vitamins, herbal and mineral supplements) within 30 days before study drug administration, or any general anaesthetic during the three months before study drug administration, and until the end of the study, with the exception of Investigator-approved hormonal contraceptives, HRT and occasional paracetamol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Bioavailability - Area under Curve of pH at 2 hours | 2 hours
  To assess the relative bioavailability of two immediate release formulations of omeprazole/sodium carbonate (Zegerid 20mg capsule and Zegerid 20mg powder for oral suspension)
Pharmacodynamics - Area under Curve of pH at 2 hours | 2 hours
  To assess the relative pharmacodynamic profiles of two immediate release formulations of omeprazole/sodium bicarbonate (Zegerid® 20mg capsule and Zegerid® 20mg powder for oral suspension).

SECONDARY OUTCOMES:
Safety and tolerability of study formulations using measurements of Cmax, tmax and t1/2 | pre-dose on day 1, and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To assess the safety and tolerability of these three formulations after single dose oral administration. To include measurements of Cmax, tmax and t1/2
Bioavailability - measurement of pH over time | 0.5, 1, 1.5, 3, 4, 8, 12, 16 and 24 hours
  To assess the relative bioavailability of an immediate release formulation of omeprazole/sodium bicarbonate (Zegerid 20mg capsule) and a delayed-release omeprazole capsule (Losec 20mg) after single dose oral administration in a fasted state. AUC of pH and % of time for pH to raise above 4 (0.5, 1, 1.5, 3, 4, 8, 12, 16 and 24 hours)
Bioavailability - measurement of pH over time | 0.5, 1, 1.5, 3, 4, 8, 12, 16 and 24 hours
  To assess the relative bioavailability of an immediate release formulation of omeprazole/sodium bicarbonate (Zegerid 20mg powder for oral suspension) and a delayed-release omeprazole capsule (Losec 20mg) after single dose oral administration in a fasted state. AUC of pH and % of time for pH to raise above 4 (0.5, 1, 1.5, 3, 4, 8, 12, 16 and 24 hours)
Pharmacodynamic Measurements of Cmax, Tmax and t1/2 | Pre-dose on day 1, and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To assess the relative pharmacodynamic profiles of an immediate release formulation of omeprazole/sodium bicarbonate (Zegerid 20mg capsule) and a delayed-release omeprazole capsule (Losec 20mg) after single dose oral administration in a fasted state.
Pharmacodynamic measurements of Cmax, Tmax and t1/2 | Pre-dose on day 1, and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To assess the relative pharmacodynamic profiles of an immediate release formulation of omeprazole/sodium bicarbonate (Zegerid 20mg powder for oral suspension) and a delayed-release omeprazole capsule (Losec 20mg) after single dose oral administration in a fasted state

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Hanna, MB BCH MRCS, Principal Investigator — Bio-Kinetic Europe, Ltd.
Locations (1):
- Bio-Kinetic Europe Limited, 14 Great Victoria Street, Belfast BT2 7BA, Belfast, United Kingdom